CLINICAL TRIAL: NCT05696392
Title: An Open-Label, Single-Arm, Phase 4 Study of Ruxolitinib Cream in Adults With Atopic Dermatitis Experiencing Sleep Disturbance in the United States (MORPHEUS)
Brief Title: The Purpose of This Study is to Evaluate the Effects of Ruxolitinib Cream on Adults With Atopic Dermatitis Experiencing Sleep Disturbance.
Acronym: MORPHEUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to lack of enrollment.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-902
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: ruoltitinib; atopic dermatitis; sleep distubance; itch; Opzelura
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group: Ruxolitinib (Experimental): ruxolitinib cream 1.5% will be applied twice daily (BID) as a thin film.
  Interventions: Drug: ruxolitinib cream

INTERVENTIONS:
Drug: ruxolitinib cream — ruxolitinib cream 1.5% will be applied twice daily as a thin film
  Other Names: INCB018424

SUMMARY:
The purpose of the study is to evaluate the effect of ruxolitinib cream on sleep disturbances with participants with Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Has clinically confirmed diagnosis of active AD according to Hanifin and Rajka (1980) criteria.
* Has at least a 2-year history of AD (information obtained from medical chart, participant's physician, or directly from the participant).
* Has an overall BSA affected by AD of 3%-20% (excluding scalp) at the screening and baseline visits.
* Has an IGA score ≥ 2 at the screening and baseline visits.
* Has an Itch NRS score ≥ 4 at the screening and baseline visits.
* Willing to complete the once-daily Itch NRS (24-hour recall period) entries at approximately the same time each day during the study.
* Agrees to maintain a regular sleep schedule during the study period.
* Willing and able to follow required study procedures for measuring sleep for the duration of the study.

Exclusion Criteria:

* Currently using a wearable or other device for monitoring sleep patterns and unwilling to discontinue its use during the study.
* Currently has a schedule that includes nighttime work shifts.
* Has had significant flares or unstable course in AD (ie, condition worsened significantly or required significant change in medications, as per medical judgment) in the previous 4 weeks before screening (information obtained from medical chart, participant's physician, or directly from the participant).
* Has received any ultraviolet B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to the screening period.
* Has had psoralen plus ultraviolet A treatment within 4 weeks prior to the screening period.
* Has received a nonbiological investigational product or device within 4 weeks prior to the screening period, or is currently enrolled in another investigational drug study.
* Has received treatment with JAK inhibitors (systemic or topical) within 4 weeks prior to the screening period.
* Has had prior treatment with a JAK inhibitor that was discontinued for safety reasons or tolerance problems.
* Has a known or suspected allergy to ruxolitinib or any component of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - First Oc Dermatology, Fountain Valley, California
  - Ark Clinical Research, Long Beach, California
  - Gw Training Center, Washington D.C., District of Columbia
  - Skin Care Research, Llc, Boca Raton, Florida
  - Driven Research Llc, Coral Gables, Florida
  - University of Florida Health Dermatology-Springhill, Gainesville, Florida
  - Skin Care Research, Llc Scr Hollywood, Hollywood, Florida
  - Ciocca Dermatology Pa, Miami, Florida
  - Trueblue Clinical Research, Tampa, Florida
  - Dermatology Specialists Research Indiana, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group Llc, Indianapolis, Indiana
  - Skin Sciences Pllc, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center (Bidmc), Boston, Massachusetts
  - Northeast Dermatology Associates, Methuen, Massachusetts
  - Essential Dermatology, Natick, Massachusetts
  - Washington University School of Medicine Dermatology, St Louis, Missouri
  - Suny Downstate Health Sciences University, Brooklyn, New York
  - Empire Dermatology, East Syracuse, New York
  - Sadick Dermatology, New York, New York
  - Skin Search of Rochester, Rochester, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Knight Cancer Institute At Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Arlington Research Center, Arlington, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Pi Coor Clinical Research Llc, Burke, Virginia
  - Clinical Research Partners Llc, Richmond, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: The purpose of this study is to evaluate the effects of ruxolitinib cream on adults with atopic dermatitis experiencing sleep disturbance. (MORPHEUS) — https://www.incyteclinicaltrials.com/study/?id=INCB%2018424-902&SearchTerm=INCB%2018424-902&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 17 study centers in the United States.
Groups:
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for up to 8 weeks to a total maximum allowed treatment area of ≤20% body surface area.
Period: Overall Study
Arm/Group | Ruxolitinib 1.5% Cream BID
Started | 47
Completed | 42
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (16.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  Black or African American | 16
  Not Reported | 1
  Captured as "Other" in Database | 1
  White | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Sleep Time (TST) as Measured by Ōura Ring Wearable Device at Week 8
Description: TST is the total amount of time spent during a planned sleep episode. Decreased TST is indicative of increased sleep disturbance. Baseline TST was the average hours of sleep within the last 7 nights prior to Visit 1. The Week 8 TST was the average hours of sleep within the last 7 nights prior to Visit 3/Week 8. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; Week 8
Population: Per Protocol Population: all participants who had no important protocol deviations. Participants must have had ≥4 nights worth of sleep data in order for the average to have been calculated; otherwise, it was set to missing. The average was based on non-missing nights of sleep data. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 11
hours
  Baseline | 5.69 (0.956)
  Change from baseline at Week 8: number analyzed (Participants) | 7
  Change from baseline at Week 8 | 0.09 (1.145)
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID; Test type: Other — difference between the average sleep at baseline and Week 8; p = 0.8357, paired t-test

2. Secondary Outcome: Change From Baseline in PROMIS Sleep Disturbance - Short Form 8b Score (24-hour Recall) at Week 8
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form 8b is a validated instrument used to measure the severity of sleep disturbance. The PROMIS score includes 8 items, each of which asks the participant to rate the severity of their sleep disturbance on a daily basis on a severity scale of 1 to 5. The PROMIS total score is calculated as the sum of the 8 items and ranges from 8 to 40. A higher PROMIS score indicates more severe sleep disturbance. The baseline score was the 7-day average of nonmissing scores for the 6 days preceding a participant's Visit 1 and their response at Visit 1. Week 8 scores comprised the 7-day average of nonmissing scores for the 6 days preceding a participant's Visit 3 and their response at Visit 3. The average was not valid and was set to missing if scores were missing on 4 or more days. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; Week 8
Population: Intent-to-Treat (ITT) Population: all participants who enrolled in the study. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 34
scores on a scale
  Baseline | 27.58 (4.955)
  Change from baseline at Week 8: number analyzed (Participants) | 24
  Change from baseline at Week 8 | -7.47 (7.802)
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID; Test type: Other — difference between the average sleep at baseline and Week 8; p = 0.0001, paired t-test

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: Adverse events have been reported for the Safety Population, comprised of all participants who received at least 1 application of study drug during the treatment period.
Arm/Group | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 7/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=47)
Application site pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to challenges with enrollment. Sample size was limited due to a high number of screen failures and important Protocol deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT05696392/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT05696392/SAP_001.pdf